CLINICAL TRIAL: NCT05305300
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Immunogenicity of a PIKA COVID-19 Vaccine in Healthy Adults Who is COVID-19 naïve or Had Previous COVID-19 Infection or Completed Inactivated or mRNA COVID-19 Vaccination.
Brief Title: A Phase I Study to Evaluate Safety, Tolerability, and Immunogenicity of a PIKA COVID-19 Vaccine in Healthy Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yisheng Biopharma (Singapore) Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: YS-009
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Vitronectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Primary Immunization (Experimental): There will be 3 dose groups, 1 to 3 with escalating antigen dose with PIKA adjuvant in sequential cohorts. A total of 45 subjects will be enrolled in Arm A. Subjects in Group 1-3 will receive two doses of PIKA COVID-19 vaccine via IM administration on Days 0 and 7.
  Interventions: Biological: PIKA COVID-19 Vaccine (CHO cell, S-protein), Arm A
- Arm B1: Booster Immunization 1 (Experimental): There will be 3 dose groups, 1 to 3 with escalating antigen dose with PIKA adjuvant in sequential cohorts. Arm B1 will enroll subjects who received Inactivated vaccines and will comprise of 15 subjects per dose. In arm B1, fifteen eligible subjects in each dose group will receive the study vaccine on Study Days 0 via intramuscular injection in alternative deltoid muscles.
  Interventions: Biological: PIKA COVID-19 Vaccine (CHO cell, S-protein), Arm B
- Arm B2: Booster Immunization 2 (Experimental): There will be 3 dose groups, 1 to 3 with escalating antigen dose with PIKA adjuvant in sequential cohorts. Arm B2 will enroll subjects who received mRNA vaccines and will comprise of 15 subjects per dose. In arm B2, fifteen eligible subjects in each dose group will receive the study vaccine on Study Days 0 via intramuscular injection in alternative deltoid muscles.
  Interventions: Biological: PIKA COVID-19 Vaccine (CHO cell, S-protein), Arm B

INTERVENTIONS:
Biological: PIKA COVID-19 Vaccine (CHO cell, S-protein), Arm A — receive two doses of PIKA COVID-19 vaccine (5 μg S protein/1mg PIKA, 10μg S protein/1mg PIKA and 20μg S protein/1mg PIKA) via IM administration on Days 0 and 7.
  Arms: Arm A: Primary Immunization
Biological: PIKA COVID-19 Vaccine (CHO cell, S-protein), Arm B — receive one dose of PIKA COVID-19 vaccine (5 μg S protein/1mg PIKA, 10μg S protein/1mg PIKA and 20μg S protein/1mg PIKA) via IM administration on Days 0.
  Arms: Arm B1: Booster Immunization 1; Arm B2: Booster Immunization 2

SUMMARY:
This is a Phase I, open label, dose-escalation study of three dose levels of the SARS-CoV-2 spike antigen administered intramuscularly (IM) in combination with a fixed dosage of PIKA adjuvant vaccine to evaluate the safety, tolerability, and immunogenicity of PIKA COVID-19 vaccine candidate in healthy individuals aged 18 years and above. The study will comprise of two arms. Arm A will include subjects who never been infected with COVID-19 or with a history of COVID-19 infection for not less than 6 months prior to study participation and Arm B will include subjects who will be receiving PIKA vaccine as a booster vaccination dose to COVID-19 primary vaccination of inactivated or mRNA Covid 19 vaccines.

DETAILED DESCRIPTION:
This is a Phase I, open label, dose-escalation study of three dose levels of the SARS-CoV-2 spike antigen administered intramuscularly (IM) in combination with a fixed dosage of PIKA adjuvant vaccine to evaluate the safety, tolerability, and immunogenicity of PIKA COVID-19 vaccine candidate in healthy individuals aged 18 years and above. The study will comprise of two arms. Arm A will include subjects who had never been infected with COVID-19 or with a history of COVID-19 infection for not less than 6 months prior to study participation and Arm B will include subjects who will be receiving PIKA vaccine as a booster vaccination dose to COVID-19 primary vaccination of inactivated or mRNA Covid 19 vaccines.

Arm A: There will be 3 dose groups, 1 to 3 with escalating antigen dose with PIKA adjuvant in sequential cohorts. A total of 45 subjects will be enrolled in Arm A. Subjects in Group 1-3 will receive two doses of PIKA COVID-19 vaccine via IM administration on Days 0 and 7. Fifteen eligible subjects in each dose group.

Arm B: There will be 3 dose groups, 1 to 3 with escalating antigen dose with PIKA adjuvant in sequential cohorts. A total of 90 subjects will be enrolled in Arm B which will be divided into Arm B1 (45 subjects) and Arm B2 (45 subjects). Arm B1 will enroll subjects who received Inactivated vaccines and will comprise of 15 subjects per dose (45 subjects). Arm B2 will enroll subjects who received mRNA vaccines and will comprise of 15 subjects per dose (45 subjects). Subjects in Group 1-3 of Arm B1 and Arm B2 will receive one booster dose of PIKA COVID-19 vaccine via IM administration on Days 0.

ELIGIBILITY:
Inclusion Criteria

Inclusion Criteria of Arm A:

1. Male and female healthy volunteers.
2. Age ≥18 years on Study Day 0.
3. Judged by the investigator to be healthy on the basis of medical history, physical examination and vital signs performed at screening.
4. Able to provide informed consent.
5. Able and willing to comply with all study procedures over follow-up period of approximately 6 months.
6. For more inclusion criteria, please contact the investigator or sponsor.

Inclusion Criteria of Arm B:

Male and female healthy volunteers.

1. Received complete primary series of COVID-19 Inactivated Vaccines not less than 6 months or Received complete primary series of COVID-19 mRNA Vaccines not less than 6 month.
2. Age ≥18 years on Study Day 0.
3. Judged by the investigator to be healthy on the basis of medical history, physical examination and vital signs performed at screening.
4. Able to provide informed consent .
5. Able and willing to comply with all study procedures over follow-up period of approximately 6 months.
6. For more inclusion criteria, please contact the investigator or sponsor.

Exclusion Criteria:

Exclusion Criteria of Arm A:

1. History of COVID-19 of less than 6 months prior to enrollment
2. Received partial or complete course of any type of COVID-19 vaccine.
3. History of close contact with a person infected or suspected of COVID-19 not less than 14 days prior to study enrollment.
4. Positive test for SARS-CoV-2 infection, including but not limited to RT-PCR /Rapid Antigen Test at screening, before the first dose (Day 0) and before the second dose (Day 7).
5. For more exclusion criteria, please contact the investigator or sponsor.

Exclusion Criteria of Arm B:

1. History of close contact with a person infected or suspected of COVID-19 not less than 14 days prior to study enrollment.
2. Positive test for SARS-CoV-2 infection, including but not limited to RT-PCR/RAT at screening, before the first dose (Day 0) .
3. Have received three and more doses of COVID-19 vaccine.
4. Pregnant or breastfeeding or intending to become pregnant or father children within the projected duration of the trial.
5. For more exclusion criteria, please contact the investigator or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Solicited local adverse events, | 7 days after each vaccination.
  Incidence of solicited local adverse events (AEs).
Solicited systemic AEs | 7 days after each vaccination.
  Incidence of solicited systemic AEs.
Unsolicited AEs | 28 days after each vaccination.
  Incidence of unsolicited AEs.
Serious adverse events (SAEs) including Suspected Unexpected Serious Adverse Reaction (SUSARs) | through study completion, an average of 6 months.
  Incidence of serious adverse events (SAEs) including Suspected Unexpected Serious Adverse Reaction (SUSARs).
Medically Attended AEs (MAAEs) | through study completion, an average of 6 months.
  Incidence of Medically Attended AEs (MAAEs).
AEs of special interest (AESIs) | through study completion, an average of 6 months.
  Incidence of AEs of special interest (AESIs).

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Liu, Ph.D, Study Director — Yisheng Biopharma CO., Ltd.
Locations (1):
- Al Kuwait Hospital (Al Baraha Hospital), Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim RJ, Qiu X, Leong RN, Gutierrez JL, Halima A, Mostafa M, Ghoneim Y, Abdrabo M, Rashad M, Hannawi S, Liu Y, Mojares Z. Safety, tolerability, and immunogenicity of PIKA-adjuvanted recombinant SARS-CoV-2 spike protein subunit vaccine in healthy adults: an open-label randomized phase I clinical trial. Clin Exp Vaccine Res. 2024 Oct;13(4):315-328. doi: 10.7774/cevr.2024.13.4.315. Epub 2024 Oct 31. PMID 39525677